CLINICAL TRIAL: NCT02822716
Title: Irreversible Electroporation for Inoperable Hepatic and Pancreatic Malignancy
Acronym: IRE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: poor case accural
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Simon Yu, Professor, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VIR-13-06
Record Dates: First submitted 2016-06-30; First posted 2016-07-04 (Estimated); Last update posted 2022-10-21 (Actual); Status verified 2022-10

CONDITIONS: Hepatic Malignant Tumors; Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Ultrasonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IRE treatment (Other): Irreversible electroporation (IRE) is a form of non-thermal local ablation for solid tumors, it induces apoptosis of tumor cells by creating irreversible damage in the cell membrane using electric current. IRE treatment is given for a therapeutic purpose as a non-surgical alternative to those patients with an inoperable condition.
  Interventions: Procedure: IRE treatment; Device: Ultrasound

INTERVENTIONS:
Procedure: IRE treatment — The treatment procedure is carried out percutaneously under ultrasound or CT guidance, or using laparoscopic or laparotomy approach when the lesion is close to hollow viscera or abdominal wall, with the patient under general anaesthesia. Insulated needle electrodes, will be placed in the treatment areas under ultrasound or CT guidance. The tumor lesion is identified, measured, and located by ultrasound or CT. Electrical current is administered in pulses with electrocardiographic synchronization to reduce the risk of cardiac arrhythmia.
Device: Ultrasound

SUMMARY:
The objectives of this study are to study the safety and effect of IRE as a treatment for inoperable hepatic and pancreatic malignancy.

DETAILED DESCRIPTION:
Irreversible electroporation (IRE) is a form of non-thermal local ablation for solid tumors, it induces apoptosis of tumor cells by creating irreversible damage in the cell membrane using electric current. The use of thermal ablation for tumors adjacent to major blood vessels is not advisable because the "heat-sink effect" owing to blood vessels render the thermal treatment not effective. On the other hand, application of thermal ablation to a tumor adjacent to blood vessels or bile ducts will cause thermal damage to these structures. It has been shown in animal experiments that IRE is effective in causing cell death while blood vessels, bile ducts, and nerves in the vicinity are preserved. Early evidence of clinical studies has shown that IRE is a reasonably safe and effective treatment for pancreatic and hepatic tumors.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for hepatic malignancy:

  1. Signed informed consent by patient
  2. Age above 18 years
  3. Child-Pugh A or B cirrhosis
  4. Eastern Cooperative Oncology Group performance (ECOG) score 2 or below
  5. No serious concurrent medical illness
  6. Histologically or cytologically proven malignant liver tumor, or lesions of size 1 to 2 cm, with typical features of hepatocellular carcinoma (HCC) on two dynamic imaging techniques, or lesions larger than 2cm, with typical features on one dynamic imaging techniques, or lesions larger than 2cm with Apha Fetal Protein (AFP) level > 200 ug/L
  7. Inoperable HCC due to patient or tumor factors, without extra-hepatic involvement on Chest X-ray (CXR) and CT
  8. Massive expansive tumor type of HCC with measurable lesion on CT
  9. Recurrent intrahepatic HCC after surgical resection or local ablation
  10. Metastatic liver tumor with well-defined margin
  11. Tumor size <= 3cm in largest dimension
  12. Tumor number <= 3
* Inclusion criteria for pancreatic malignancy:

  1. Signed informed consent by patient
  2. Age older than 18 years.
  3. Any kind of histologically or radiologically diagnosed malignant pancreatic tumor.
  4. Tumor size <= 3cm in largest dimension
  5. Surgical treatment is considered not an option because of patient factors or tumor factors, such as those with vascular encasement or regional lymph node metastasis
  6. Locally recurrent pancreatic tumor after surgical resection
  7. Karnofsky's performance status of 50% or greater.
  8. Life expectancy greater than 3 months.
  9. Normal coagulation profile (INR <1.5; platelet count >50 10^9/L).
  10. Willingness and ability to complete follow-up interviews and imaging investigations following the treatment.

Exclusion Criteria:

* Exclusion criteria for hepatic malignancy:

  1. History of prior malignancy except on the condition that the patient has been disease free for ≥3 years
  2. Concurrent ischemic heart disease or heart failure
  3. Biliary obstruction not amenable to percutaneous drainage
  4. Child-Pugh C cirrhosis
  5. Intractable ascites not controllable by medical therapy
  6. History of variceal bleeding within last 3 months; serum total bilirubin level > 50 umol/L
  7. Serum albumin level < 25g/L
  8. INR > 1.5, platelet count <50 10^9/L
  9. Infiltrative or diffuse tumor
  10. Hepatic vein tumor thrombus
  11. Pregnancy
  12. Cardiac arrhythmia
  13. Uncontrolled hypertension
* Exclusion Criteria for pancreatic malignancy:

  1. Patient has active infection.
  2. Patient has bleeding tendency.
  3. Presence of portal vein thrombus.
  4. Tumour size of greatest dimension >3cm.
  5. Tumor with ill defined infiltrative margin.
  6. The tumor has invaded the duodenal wall.
  7. Presence of distant metastasis
  8. Currently experiencing an episode of major mental illness (psychosis, major affective disorder, or schizophrenia).
  9. Pregnancy
  10. Cardiac arrhythmia
  11. Uncontrolled hypertension

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2013-07-22 (Actual); Primary Completion 2020-09-23 (Actual); Study Completion 2020-09-23 (Actual)

PRIMARY OUTCOMES:
Radiological assessment | 1 month
  CT scan will be performed. Tumor response will be assessed using RECIST criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Simon Yu, Professor, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Department of Imaging and Interventional Radiology, Prince of Wales Hospital, The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No